CLINICAL TRIAL: NCT05460728
Title: Dry Needling Effects on Spasticity and General Functioning in Patients With Traumatic Brain Injury: A Case Study
Brief Title: Dry Needling Effects Post-traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anas Radi Hassan Alashram (Other)
Responsible Party: Sponsor-Investigator, Anas Radi Hassan Alashram, Associate Professor, Middle East University
Organization: Middle East University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SREC/22/05/041
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry needling (Experimental)
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling — A three-weekly session of DNT was administered with an acupuncture needle (0.30 × 50 mm; Huan Qiu, Suzhou, China). For each session, DNT was applied in the deltoid, biceps brachialis, wrist extensors and flexors, thenar muscles, vastus medialis, gastrocnemius medialis, and tibialis anterior (Hong, 1994). Following focal twitch responses (maximum three), the dry needle was left inserted for 15 minutes in each muscle.

SUMMARY:
Thirty-six years old male with a history of TBI with compromised functionality of the right upper and lower limbs, spasticity, distributed balance, and difficulties performing independent gait has participated in the study. Berg balance scale, 6-minute walk test, modified Ashworth scale, and functional independence measure was used to assess balance, gait, spasticity, and functional intemperance, respectively.

DETAILED DESCRIPTION:
A 36-year-old man (height: 1.75 m, weight: 73 kg) with a 6-month history of TBI due to a motor vehicle accident resulting in right hemiplegia was admitted in March 2022 to the outpatient Neurological Physiotherapy Clinic. He was alert and oriented and had expressive aphasia. The patient had compromised functionality of the right upper and lower limbs, spasticity, distributed balance, and difficulties performing independent gait. He was right-hand dominant.

Demographic data were recorded including age, gender, occupation, and duration of disease. The outcome measures were evaluated at baseline (T0), 12 weeks from T0 (T1), and 16 weeks from T0 (4 weeks after the intervention, T2).

Spasticity assessment Spasticity for the upper and lower limbs was evaluated using the modified Ashworth Scale (MAS). The scale evaluates the resistance of a limb to a rapid passive stretch in 6 scores from 0 to 5. Score 0 indicates normal muscle tone, and 5 indicates rigid limb. The MAS for a patient with TBI has shown good reliability (ICC = 0.62-0.90).

Gait and balance assessment The primary outcome of the 6-MWT was the distance covered by the patient in 6 minutes. It was used to evaluate functional capacity in individuals with chronic disorders. The 6-MWT is a good predictor of cardiorespiratory endurance in patients with TBI. The 6-MWT for a patient with TBI has shown good reliability (ICC = 0.96-0.98) and good discriminant validity. The test was applied according to the guidelines provided by of American Thoracic Society (ATS). Two reference points were placed at 30 m from each other. Before and immediately following the test, heart rate and oxygen saturation were taken using a pulse oximeter. The patient was able to complete the 6-MWT without taking a rest break. Gait speed was demonstrated in meters per minute by dividing the total distance covered in the 6-MWT by 6 minutes.

The balance and risk of falls were evaluated using Berg Balance Scale (BBS). This scale includes 14 items requiring patients to complete tasks related to the everyday life of varying difficulty levels. The total final scores range from 0 to 56. A total score of fewer than 45 exhibits balance impairment. The BBS has excellent reliability (ICC = 0.986) in patients with TBI.

Independence measure The Functional Independence Measure (FIM) is a tool that measures the individual's degree of dependency. Thirteen tasks belong to a motor and 5 to a cognitive element. Each activity is evaluated on a 7-point scale ranging from 1 (complete dependency) to 7 (complete autonomy). A total scores range from 18 to 126, corresponding to 13-91 for the motor subscore and 5-35 for the cognitive sub-score.

Intervention The intervention was performed in an outpatient Neurological Physiotherapy Clinic, Amman, Jordan, by a skilled physical therapist. The MTrPs were detected in the upper and lower limbs based on the DNT criteria for spasticity: 1) Fundamental criteria: Limitation to passive stretching or activating of myotatic reflex and tight muscle band, and 2) Affirmative criteria: visual or tactile identification of global or focal twitch response when inserting the needle, and neural release (i.e. immediate release from contraction).

A three-weekly session of DNT was administered with an acupuncture needle (0.30 × 50 mm; Huan Qiu, Suzhou, China). For each session, DNT was applied in the deltoid, biceps brachialis, wrist extensors and flexors, thenar muscles, vastus medialis, gastrocnemius medialis, and tibialis anterior. Following focal twitch responses (maximum three), the dry needle was left inserted for 15 minutes in each muscle.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury

Exclusion Criteria:

* Unstable status

Ages: 30 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-09 (Actual)

PRIMARY OUTCOMES:
modified Ashworth Scale (MAS) | Change from baseline MAS at 12-week and 16-week
  Spasticity for the upper and lower limbs was evaluated using the modified Ashworth Scale (MAS) (Ghotbi, 2009). The scale evaluates the resistance of a limb to a rapid passive stretch in 6 scores from 0 to 5. Score 0 indicates normal muscle tone, and 5 indicates rigid limb (Bohannon, 1987). The MAS for a patient with TBI has shown good reliability (ICC = 0.62-0.90) (Mehrholz, 2005).

SECONDARY OUTCOMES:
6-Minute Walk Teat (6-MWT) | Change from baseline 6-MWT at 12-week and 16-week
  The 6-Minute Walk Teat (6-MWT) was the distance covered by the patient in 6 minutes. It was used to evaluate functional capacity in individuals with chronic disorders (Danielsson, 2007). The 6-MWT is a good predictor of cardiorespiratory endurance in patients with TBI (Mossberg, 2012). The 6-MWT for a patient with TBI has shown good reliability (ICC = 0.96-0.98) and good discriminant validity (Bartels, 2012). The test was applied according to the guidelines provided by of American Thoracic Society (ATS) (ATS Statement,2002). Two reference points were placed at 30 m from each other. Before and immediately following the test, heart rate and oxygen saturation were taken using a pulse oximeter. The patient was able to complete the 6-MWT without taking a rest break. Gait speed was demonstrated in meters per minute by dividing the total distance covered in the 6-MWT by 6 minutes.
Berg Balance Scale (BBS) | Change from baseline BBS at 12-week and 16-week
  The balance and risk of falls were evaluated using Berg Balance Scale (BBS). This scale includes 14 items requiring patients to complete tasks related to the everyday life of varying difficulty levels. The total final scores range from 0 to 56. A total score of fewer than 45 exhibits balance impairment (Berg,1989; Zwick,2000). The BBS has excellent reliability (ICC = 0.986) in patients with TBI (Newstead,2005).
Functional Independence Measure (FIM) | Change from baseline FIM at 12-week and 16-week
  The Functional Independence Measure (FIM) is a tool that measures the individual's degree of dependency. Thirteen tasks belong to a motor and 5 to a cognitive element. Each activity is evaluated on a 7-point scale ranging from 1 (complete dependency) to 7 (complete autonomy). A total scores range from 18 to 126, corresponding to 13-91 for the motor subscore and 5-35 for the cognitive sub-score (Hamilton, 1987).

CONTACTS AND LOCATIONS:
Overall Officials: ANAS RADI H Annino, Study Director — University of Rome Tor Vergata
Locations (1):
- Isra University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No